CLINICAL TRIAL: NCT00669968
Title: PET Myocardial Perfusion Imaging With CT Angiography and Measurement of Coronary Flow Reserve: A Prospective Study of Effectiveness, Impact on Patient Management, Prognostic Value, and Downstream Costs
Brief Title: Study of Value of Cardiac PET Scans With or Without CT Angiography and/or Measurement of Coronary Flow Reserve
Status: Completed | Type: Observational
Sponsor: Kettering Health Network (Other)
Responsible Party: Sponsor
Other Study IDs: 07-034
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Chest Pain; Coronary Artery Disease
Keywords: PET myocardial perfusion imaging; Cardiac PET; Rubidium; Coronary Artery CT Angiogram; Coronary Flow Reserve; Adenosine stress test
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
How does PET myocardial perfusion imaging involving CT angiography and measurement of coronary flow reserve affect patient care.

DETAILED DESCRIPTION:
The purpose of this research is to determine how PET myocardial perfusion imaging involving CT angiography and measurement of coronary flow reserve affects patient care. This research will also compare the effectiveness of these scans to other similar tests and compare the cost-effectiveness of these scans to other similar tests over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to Kettering Medical Center for PET myocardial perfusion imaging with or without CTA and/or coronary flow reserve measurement.
* Patients over 18 years of age.

Exclusion Criteria:

* Patients who do not consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo Rubidium PET adenosine stress test with or without CT angiography of coronary arteries and/or coronary flow reserve measurment at Kettering Medical Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Dittoe, MD, Principal Investigator — Kettering Health Network
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States